CLINICAL TRIAL: NCT05248477
Title: Improve the Survival Without Morbidity of Extremely Preterm Infants: A Stepped-wedge Cluster-randomized Trial
Brief Title: Improve the Survival Without Morbidity of Extremely Preterm Infants (PREMEX)
Acronym: PREMEX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: APHP211004; 2021-A02520-41 (Other: ID-RCB Number)
Record Dates: First submitted 2021-12-20; First posted 2022-02-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Newborn; Extreme Prematurity; Pretrm Infants
Keywords: extremely preterm infants; periviable birth; perinatal management; EXPRIM protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual practice (No Intervention)
- Premex protocol (Experimental): a new organization of care, based on the EXPRIM (EXtrem PRematurity Innovative Management) protocol, involving early, standardized, and multidisciplinary management of women hospitalized for a risk of extremely preterm birth and their children
  Interventions: Other: Premex Protocol

INTERVENTIONS:
Other: Premex Protocol — This protocol presupposes stages during which staff are informed and trained. It is based on the following principles:
  * Administration of corticosteroid therapy to all eligible women, independent of the decision about active or palliative care
  * A prognostic evaluation in a non-emergency meeting of the obstetricians and neonatologists/pediatricians involved, no longer based only on gestational age, and enabling the team to provide consistent, consensual, and individualized information to parents;
  * A joint decision about the obstetric and neonatal (active or palliative) care to be proposed to parents at the end of this evaluation;
  * An interview with parents, also on non-emergency basis, to give them information about the child's prognosis and the management proposed, to answer their questions, and to obtain their opinion;
  * Management at birth consistent with that decided in consultation with the parents.
  Arms: Premex protocol

SUMMARY:
The intervention proposed is a new organization of care, based on the EXPRIM (EXtrem PRematurity Innovative Management) protocol, involving early, standardized, and multidisciplinary management of women hospitalized for a risk of extremely preterm birth and their children. It will take place in each perinatal network for all pregnant women hospitalized between 22 and 26 weeks with a risk of preterm delivery.

Setting up the protocol requires taking into account the parents' time and timing issues, and its potential for change, to plan the implementation of the protocol, especially the degree of emergency of the situation and the probability of imminent delivery.

The follow-up collected for this study will take place:

* At D4 post-delivery: A questionnaire about the parents' experience of the information delivered and the decisions made will be given to and collected from the parents
* At Day 28, post-delivery: A questionnaire about the parents' experience of care for their child will be given to and collected from the mother and the co-parent.
* At the child's discharge from the hospital, or if he or she dies in the hospital:

  * Collection of clinical data (principal endpoint) from data in the medical file.
  * Data to measure practices and adherence to the intervention will be collected
* When the child reaches the corrected age of 2 years:

  * a short questionnaire will be completed by the physician caring for the child at the corrected age of 2 years. The data collected will concern motor and sensory development, in particular, cerebral palsy, blindness, and deafness..
  * Information about the child's development will also be collected with a questionnaire including a standardized assessment scale, he PARCA-R questionnaire (Parent Report of Children's Abilities-Revides), which the parents will complete.

DETAILED DESCRIPTION:
Extremely preterm infants, those born between 22 and 26 weeks of gestation, are at very high risk of neonatal death, severe morbidity, and disabilities. These children's survival basically depends on the obstetric-pediatric team's willingness to provide active care. In France, practices vary strongly according to the child's place of birth. The rates of active antenatal care (reflects the intention to manage the child actively at birth), standardized by gestational age, vary from 22% to 61% between regions. One of the consequences of this heterogeneity is that the survival rate in France of these extremely premature infants is much lower than that of countries offering similar levels of care. Among the children live-born in France, survival rates at hospital discharge were 0% at 22 weeks, 1% at 23, 31% at 24, 59% at 25, and 75% at 26 weeks. Survival in the USA, Great Britain, Japan, Australia, and Sweden ranges from 10 to 50% higher than in France.

The great variability of antenatal practices for the management of extremely preterm infants reflects the disarray of medical teams. In the absence of consensus and written decision-making processes, this uncertainty culminates in management decisions based at best on local habits and at worst on the individual habits of the clinician present. These habits vary with the physicians' beliefs or convictions, and their level of knowledge and experience of extremely preterm births. This variability of practices between hospitals presents a problem of equity.

The hypothesis is that standardization of the management of extremely preterm infants, from the moment that the pregnant woman is hospitalized until the child's birth should improve survival without severe morbidity in this group of children at very high risk

The intervention proposed is a new organization of care, based on the EXPRIM (EXtrem PRematurity Innovative Management) protocol (MC Lamau, et al, PMID: 34059380), involving early, standardized, and multidisciplinary management of women hospitalized for a risk of extremely preterm birth and their children. It will take place in each perinatal network for all pregnant women hospitalized between 22 and 26 weeks with a risk of preterm delivery.

Setting up the protocol requires taking into account the parents' time and timing issues, and its potential for change, to plan the implementation of the protocol, especially the degree of emergency of the situation and the probability of imminent delivery.

Complex intervention, named the EXPRIM protocol, aimed at standardizing the organization of care. It is based on the following principles:

* A collective obstetric-pediatric prognostic assessment, in a non-emergency setting, no longer based only on gestational age, and ensuring better team consistency in terms of the attitude to propose to parents;
* A consensus decision by the multidisciplinary team about the obstetric and neonatal management proposed-either active or palliative care-at the conclusion of this prognostic evaluation
* An interview with the parents to:

  * inform them about the obstetric situation and the child's prognosis
  * answer their questions
  * propose either active or palliative care to them as management
  * and then ask their opinion.
* The administration of corticosteroid therapy, independently of the decision about management (active or palliative care), starting at 23 weeks will be of broad indication;

If the hospitalization takes place in a level-1 or 2 hospital: after general information about preterm delivery, a proposal to transfer the woman to the perinatal network's level-3 hospital, starting at 23 weeks

The choice of a stepped-wedge cluster randomization design allows all perinatal networks to implement the intervention.

After the random drawing of clusters for the intervention, the teams will be trained in the EXPRIM protocol and then will undergo a 3-month transition period (not considered either a control or intervention period) to learn the protocol thoroughly. The data collected during this period will not be used in the analysis. In summary, the 3 stages before recruitment during the intervention are:

1. allocation of clusters
2. training of perinatal teams
3. transition period After random drawing, 4 perinatal networks will be allocated to the intervention in 5 waves every 3 months, with 3 months of recruitment for the last wave. Twenty perinatal networks will be randomized and will participate in the trial with a total recruitment period of 21 months (including the 3-month transition periods). Overall, the duration of the study at each center will be 49 months. All perinatal networks will have a period with and without the intervention and will participate in the comparison accordingly. After 15 months all the networks will have begun the intervention.

No specific follow-up visit for the purposes of the study is planned. The hospital staff physicians will perform follow-up as part of the standard usual care for women and their newborns.

The follow-up collected for this study will take place:

* At D4 post-delivery (or before, if the woman leaves the hospital before then): A questionnaire about the parents' experience of the information delivered and the decisions made will be given to and collected from the parents. There are 2 "parental experience" questionnaires: one destined to parents of newborn alive and admitted in NICU and one destined to parents of stillborn or deceased child at birth. For parents of a stillborn or deceased child at birth, this questionnaire may be given during hospitalization in maternity (D0-D4), or after returning home or during the postnatal visit.
* At Day 28, post-delivery: A "Neonatal individualized developmental care questionnaire about the parents' experience of care for their child will be given to and collected from the mother and the co-parent.
* At the child's discharge from the hospital, or if he or she dies in the hospital:

  * Collection of clinical data (principal endpoint) from data in the medical file. If the patient was transferred to another hospital, the PREMEX investigator and/or the CRT will obtain the follow-up data to enter on the e-CRF.
  * Data to measure practices and adherence to the intervention will be collected
  * The neonatologist-investigator will ask the parents at the child's discharge from hospitalization for written consent to continue their participation in this study for the follow-up at age 2.
* When the child reaches the corrected age of 2 years:

  * Nearly all the surviving children will be receiving care within structured networks for the follow-up of vulnerable children, responsible for optimizing their medical care and follow-up. Accordingly, a short questionnaire will be completed by the physician caring for the child at the corrected age of 2 years. The data collected will concern motor and sensory development, in particular, cerebral palsy, blindness, and deafness. The questionnaire will be sent to the parents, who will ask the physician to complete it at the medical visit planned at this age. The physician will send the completed questionnaire to the project coordinators.
  * Information about the child's development will also be collected with a questionnaire including a standardized assessment scale, the PARCA-R questionnaire (PArent Report of Children's Abilities-Revised). Parents will be invited to complete the PRO (Patient Reported Outcomes, the PARCA-R questionnaire in our case) on an electronic platform-Patient Reported Outcomes-and will receive specific access codes.

At the time of inclusion, the contact data of the parents taking part in the study (e-mail address, telephone number and postal address) were collected on contact forms by the clinical teams of each maternity unit and kept in the medical files.

As part of the 2-year follow-up of these children, the coordinating midwife and/or CRT centralized will collect this contact data from the maternity units via a secure.

ELIGIBILITY:
Inclusion Criteria:

Mothers:

* women hospitalized between 22 and 26 weeks for risk of preterm delivery with a fetus alive or dead at admission and with a delivery between 22 and 26 completed weeks
* understanding of the French language by the woman or in the immediate entourage in charge of the child.

Children: all newborns (live- and stillborn) delivered between 22 and 26 weeks.

Exclusion Criteria

* women who object to the use of their routine perinatal data,
* women giving birth before 22 weeks and after 26 completed weeks.
* woman to legal protection (subject protected by law under guardianship or curatorship)
* Women undergoing a termination of pregnancy (TOP) for severe congenital anomaly or psycho-social contexte

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2377 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
survival at hospital discharge without severe morbidity (composite outcome) | Up to 24 Weeks
  Severe morbidity is a composite criterion assessed up to 40 post-menstrual age (PMA) and defined by at least one of the following severe neonatal morbidities:
  * Severe bronchopulmonary dysplasia, defined by the need for oxygen therapy and/or mechanical ventilatory support (endotracheal or noninvasive) at 36 weeks PMA (Jobe 2001).
  * Severe intraventricular hemorrhage (IVH), defined by IVH of either grade 3, associated with ventricular dilation, or grade 4, which is associated with a hemorrhagic lesion of the adjacent parenchyma) (Volpe 2009).
  * Severe retinopathy, defined as retinopathy of prematurity (ROP) of type 3 or higher according to the international classification (ICCROP 2005) and/or need for laser treatment.
  * Severe enterocolitis, defined as types 2 and 3 in the modified Bell's classification (Bell, 1978).
  * Periventricular leukomalacia, defined by cavities in the periventricular white matter on ultrasound.

SECONDARY OUTCOMES:
Child's survival at hospital discharge | Up to 24 Weeks
  Number of living children
Neurosensory condition ( composite outcome) | at a corrected age of 2 years.
  Neurosensory condition, assessed by the pediatrician responsible for monitoring the child
  * cerebral palsy, defined by the European classification (European Cerebral Palsy Network 2000) as any permanent motor deficiency resulting from a nonprogressive lesion of the immature brain. This term makes it possible to cover all motor impairments. The severity of the motor impairment will be assessed by the 5-level international GMFCS (classification system of gross motor function, Ghassabian 2016): the child walks w/o limitations (level 1), walks w/ limitations (level 2), walks using a handheld mobility device (level 3), has self-mobility w/ limitations (level 4), is transported in a manual wheelchair (level 5). Cerebral palsies of level 1 are minor, those of level 2 moderate, and those of levels 3-5 severe;
  * visual deficiency is defined by unilateral (moderate) or bilateral (severe) blindness
  * auditory deficiency is defined by unilateral (moderate) or bilateral (severe) deafness
child's global development | at a corrected age of 2 years.
  Assessment of the child's global development will be based on a standardized parent-completed questionnaire: the PArent Report of Children's Abilities-Revised (PARCA-R). This questionnaire is a validated parent report instrument measuring the child's non-verbal cognition (communication, gross motor skills, fine motor skills, problem resolution, and social relations). This questionnaire includes a series of 34 questions and is valid over a four-month window from 23.5 to 27.5 months of corrected age. The questionnaire has been age-standardised and results are provided in percentiles relative to norms in the term population.
Medical economics: | at a corrected age of 2 years
  Incremental cost-effectiveness ratio (ICER) defined by the ratio of the cost difference from the hospital's oint of view to the difference in survival, both overall and without severe morbidity; budgetary impact, assuming the widespread dissemination of these practices throughout France.
Parents' experience of the information they received, their involvement in decision making, and the decisions made | on day 4
  This experience will be assessed by 10 simple questions to obtain responses on a scale ranging from 0 ("No, not at all") to 10 ("Yes, agree completely").
Parents' implication in Neonatal individualized developmental care | on day 28
  This experience will be assessed by 10 simple questions to obtain responses on a scale ranging from 0 ("No, not at all") to 10 ("Yes, agree completely").

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Henri JARREAU, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Pierre-Yves ANCEL, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lamau MC, Ruiz E, Merrer J, Sibiude J, Huon C, Lepercq J, Goffinet F, Jarreau PH. A new individualized prognostic approach to the management of women at risk of extreme preterm birth in France: Effect on neonatal outcome. Arch Pediatr. 2021 Jul;28(5):366-373. doi: 10.1016/j.arcped.2021.04.005. Epub 2021 May 28. PMID 34059380